CLINICAL TRIAL: NCT03403452
Title: A Exploratory Clinical Trial Study on Apatinib in the Treatment of Metastatic Colorectal Cancer Who Have Progressed After Standard Second Line Therapy
Brief Title: Apatinib in the Treatment of Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xu jianmin, Director of colorectal surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APAMCRC
Record Dates: First submitted 2018-01-06; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm for Apatinib (Experimental): 500 mg,p.o.,qd
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 500 mg,p.o.,qd, until disease progression or intolerable toxicity or patients withdrawal of consent.

SUMMARY:
This is an Exploratory Clinical Trial Study on Apatinib in the Treatment of Metastatic Colorectal Cancer Who Have Progressed after Standard Second Line Therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 80 years of age
* Histological confirmed advanced or metastatic colorectal cancer，at least one measurable lesion, larger than 10 mm in diameter by spiral CT
* Have failed for ≥ 2 lines of chemotherapy and/or targeted therapy
* Life expectancy of more than 3 months
* ECOG performance scale 0～1
* Duration from the last therapy is more than 4 weeks for operation, radiotherapy or cytotoxic agents
* Adequate hepatic, renal, heart, and hematologic functions (platelets > 80 ×10^9/L, neutrophil > 1.5 × 10^9/L, serum creatinine ≤ 1×upper limit of normal(ULN), bilirubin < 1.5 ULN, and serum transaminase ≤ 2.0× ULN)
* Child bearing potential, a negative urine or serum pregnancy test result before initiating apatinib, must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article. Male: All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study and for 8 weeks after the last dose of test article.
* Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Prior VEGFR inhibitor treatment within 2 weeks
* History of other malignancies within 5 years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Preexisting uncontrolled hypertension defined as more than 140/90 mmHg despite using single medical therapy
* More than class I (NCI CTCAE 3.0 ) myocardial ischemia, arrhythmia(including QTcF:male ≥ 450 ms, female ≥ 470 ms), or cardiac insufficiency myocardial ischemia, arrhythmia, or cardiac insufficiency
* Pregnant or lactating women
* Before or at the same time any, second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* URT: urine protein ≥ (++)and > 1.0 g of 24 h
* PT, APTT, TT, Fbg abnormal, having hemorrhagic tendency or receiving the therapy of thrombolysis or anticoagulation
* Certain possibility of gastric or intestine hemorrhage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS（progress free survival） | From assignment of the first subject to 3 months later after the last participant is recruited
  PFS was defined as the time from assignment to disease progression radiological/clinical or death due to any cause

SECONDARY OUTCOMES:
OS（overall survival） | From assignment of the first subject until 30 death events observed, up to 2 years
  OS is defined as the time from date of assignment to death due to any cause
ORR（objective response rate） | From assignment of the first subject to 3 months later after the last participant is recruited
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)
DCR（disease control rate) | From assignment of the first subject to 3 months later after the last participant is recruited
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No